CLINICAL TRIAL: NCT05512273
Title: Evaluation of Implant Site Preparation With Piezosurgery vs Conventional Drills in Terms of Operation Time, Implant Stability and Bone Density. (Randomized Controlled Clinical Trial- Split Mouth Design)
Brief Title: Implant Site Preparation With Piezosurgery vs Conventional Drills in Terms of Operation Time, Implant Stability and Bone Density
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Piezosurgery_22
Record Dates: First submitted 2022-08-17; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Implant Osteotomy

STUDY DESIGN:
Intervention Model Description: Split mouth
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study (Experimental)
  Interventions: Procedure: Piezosurgery assisted osteotomy
- Control (Active Comparator)
  Interventions: Procedure: Conventional drilling osteotomy

INTERVENTIONS:
Procedure: Piezosurgery assisted osteotomy — Sequential osteotomy drilling was done using mectron piezosurgery implant drilling protocol
  Arms: Study
Procedure: Conventional drilling osteotomy — bone osteotomy for implant placement was done following the BEGO Semados RS/RSX TrayPlus conventional drilling
  Arms: Control

SUMMARY:
The preparation of the implant site has a major influence on the success rate and long-term survival of dental implants. Piezoelectric devices and special implant drilling inserts are now emerging to replace conventional drills.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bilateral missing premolars
* Remaining bone height more ≥ 10mm.
* Remaining bone width ≥ 6mm

Exclusion Criteria:

* patients that smoke more than 10 cigarettes/day
* Patients with uncontrolled systemic disease.
* Presence of bone pathology within the future osteotomy site

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Time of surgery | through operation completion
  Average surgical times for implant site was estimated
Change in implant stability | at baseline and 4 months
  ISQ was measured using ostell device
Change in bone density | at baseline and 4 months
  Mean bone density using CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Beirut Arab University, Beirut, Lebanon

REFERENCES:
- [Derived] Arakji H, Osman E, Aboelsaad N, Shokry M. Evaluation of implant site preparation with piezosurgery versus conventional drills in terms of operation time, implant stability and bone density (randomized controlled clinical trial- split mouth design). BMC Oral Health. 2022 Dec 3;22(1):567. doi: 10.1186/s12903-022-02613-4. PMID 36463145